CLINICAL TRIAL: NCT00796770
Title: Vaccination of HIV-1 Infected Patients With Ex-vivo Generated Interferon-α Dendritic Cells Loaded With HIV-1 Lipopeptides and Activated With Lipopolysaccharide in Addition to Antiretroviral Treatment: Exploratory Phase I Study-(DALIA Trial)
Brief Title: Vaccination of HIV-1 Infected Patients With Dendritic Cells in Addition to Antiretroviral Treatment - (DALIA Trial)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 008-017
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: HIV
Keywords: HIV; Vaccine; HAART; HIV-1; AIDS; Dendritic Cells; DALIA
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dendritic Cell Vaccine (Experimental): Autologous dendritic cells generated using GM-CSF and interferon alpha, loaded with HIV lipopeptides and activated with lipopolysaccharide
  Interventions: Biological: Dendritic Cell Vaccine

INTERVENTIONS:
Biological: Dendritic Cell Vaccine — Biological/Vaccine: Experimental: Dendritic Cell Vaccine Patients will receive 4 doses of the vaccine at weeks 0, 4, 8 and 12. The vaccine will be injected subcutaneously, in 3 separate injection sites in the upper and lower extremities.
  At week 24, patients will have HAART treatment interrupted. The HAART treatment will be resumed at week 48 or earlier at any time point if one of the following occur:
  1. two consecutive measurements of CD4+ T cell count below 350x10e6 cells/L and/or 25% of total lymphocytes within at least a 2 weeks
  2. an opportunistic infection
  3. a CDC class C-defining event (defined in appendix 2)
  4. a serious non-AIDS defining event.
  Patients will have follow-up visits on weeks: 22, 24, 25, 26, 27, 28, 32, 36, 40, 44, and 48.

SUMMARY:
The purpose of this study is to determine whether the administration of a dendritic cell vaccine is a safe and effective treatment for HIV-1 patients.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the administration of a dendritic cell vaccine is a safe and effective treatment for HIV-1 patients. This will be a phase I, single-center, study in HIV infected patients. The primary objective is to evaluate safety of the vaccination schedule (from apheresis procedure to week 24) at week 24 and safety of the Analytical Treatment Interruption (ATI; from week 24 to week 48) at week 48 in HIV-1 infected patients who have been receiving antiretroviral therapy for at least 12 months with HIV-1 RNA ≤50 copies/mL and CD4+ T cell counts >500/mm3 at entry in the trial and who received, in addition to anti-retroviral therapy for 24 weeks, vaccination with ex vivo generated interferon-alpha dendritic cells loaded with HIV-1 lipopeptides and activated with lipopolysaccharide (BIIR/ANRS-HIVax-001, the DC vaccine product).

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old
2. written informed consent
3. HIV1 infection documented by any licensed ELISA test kit and confirmed by Western Blot at anytime prior to study entry
4. on treatment with a combination of antiviral drugs (HAART) for at least 12 months, and stable on treatment for at least 3 months prior to enrollment. HAART is defined as an antiretroviral regimen consisting of at least three registered antiretroviral drugs (other than 3 Nucs only and low dose ritonavir used for boosting other protease inhibitors does not count as one of these three antiretroviral agents)
5. CD4+ T cell counts > 500 cells/mm3 on at least two consecutive measurements (including the screening value) within the previous 6 months prior to enrollment (occasional CD4 cell counts ranging between 450-500 cells/mm3 is permitted)
6. nadir CD4+ T cell counts > 300 cells/mm3 prior HAART
7. plasma HIV-RNA ≤ 50 copies/mL on at least two consecutive measurements (including the screening value) within the previous 3 months prior to enrollment (occasional so called 'blips' up to 200 copies/mL are permitted)
8. no history of CDC class C event (Appendix 2)
9. no vaccination in the last 3 months
10. blood cells and chemistry:

    1. neutrophils ≥ 1,000/mm3
    2. platelets ≥ 100,000/mm3
    3. hemoglobin ≥ 10 g/dl
    4. creatinin ≤ 1.5 x N
    5. ASAT, ALAT, conjugated bilirubin ≤ 2.5 x N
11. Adequate Kidney Function proteinuria ≤ 1 g/l (++)by urinalysis

Exclusion Criteria:

1. Nadir CD4+ T cell counts < 300 cells/mm3 prior HAART
2. pregnant or lactating woman
3. any prior chemotherapy treatment
4. interferon alpha (IFN-α-2b) or sargramostim (GM-CSF) < 12 weeks before the beginning of the trial
5. interleukin-2 (IL-2) <12 weeks before the beginning of the trial,
6. corticosteroids or other immunosuppressive agents <12 weeks before beginning the trial
7. active asthma and/or on treatment for asthma,
8. any history of malignancy (except basal carcinoma of the skin) including any hematologic malignancy or AIDS defining malignancy, such as lymphoproliferative disorder or Kaposi's sarcoma. Patients with Kaposi's sarcoma limited to the skin that disappeared while on HAART therapy, and without requiring any other systemic therapy, 1 year prior to study entry will be eligible to participate
9. angina pectoris or with congestive heart failure, with auto-immune disease, or evolutive pulmonary disease, or organ failure
10. active infections including viral hepatitis
11. history of thrombocytopenia
12. chronic hepatitis B or C
13. previous exposure to any HIV experimental vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of the vaccination schedule at week 24 and the safety of the Analytical Treatment Interruption at week 48 in HIV-1 infected patients. | May 2010

SECONDARY OUTCOMES:
To evaluate immune responses using several defined assays as well as viral and CD4+ T cell status | May 2010

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Banchereau, PhD, Principal Investigator — Baylor Research Institute
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Alexandre M, Prague M, Lhomme E, Lelievre JD, Wittkop L, Richert L, Levy Y, Thiebaut R. Definition of Virological Endpoints Improving the Design of HIV Cure Strategies Using Analytical Antiretroviral Treatment Interruption. Clin Infect Dis. 2024 Dec 17;79(6):1447-1457. doi: 10.1093/cid/ciae235. PMID 38819800
- [Derived] Cobb A, Roberts LK, Palucka AK, Mead H, Montes M, Ranganathan R, Burkeholder S, Finholt JP, Blankenship D, King B, Sloan L, Harrod AC, Levy Y, Banchereau J. Development of a HIV-1 lipopeptide antigen pulsed therapeutic dendritic cell vaccine. J Immunol Methods. 2011 Feb 28;365(1-2):27-37. doi: 10.1016/j.jim.2010.11.002. Epub 2010 Nov 18. PMID 21093448